CLINICAL TRIAL: NCT07264439
Title: Evaluation of the Effectiveness of Virtual Reality Headsets With Hypnotic Scenarios for Hygiene Care in Patients With Alzheimer's Disease or Related Disorders (ADRD) With Behavioral Disturbances
Brief Title: Evaluation of the Effectiveness of Virtual Reality Headsets With Hypnotic Scenarios for Hygiene Care in Patients With Alzheimer's Disease or Related Disorders With Behavioral Disturbances
Acronym: HYPNOGER 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0010
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Effectiveness; Virtual Reality; Hypnotic Scenarios; Hygiene Care; Alzheimer's Disease and Related Disorders (ADRD); Behavioral Disturbances
Keywords: Effectiveness; virtual reality; hypnotic scenarios; hygiene care; Alzheimer's disease and related disorders (ADRD); behavioral disturbances
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled trial (Active Comparator)
  Interventions: Other: standard cares
- VR headset (Experimental): a virtual reality (VR) headset with hypnotic scenarios
  Interventions: Device: VR headset

INTERVENTIONS:
Device: VR headset — VR headset enabling the management of hypnotic scenarios. The headset will project immersive 3D images and deliver a hypnotic narrative, thus combining VR and hypnosis-based techniques. This intervention will be applied during hygiene and toileting care and compared to standard behavioral management traditionally used in the structures.
  Arms: VR headset
Other: standard cares — standard cares
  Arms: controlled trial

SUMMARY:
A device combining a virtual reality (VR) headset with hypnotic scenarios may represent an effective tool to reduce anxiety and opposition during hygiene care in patients with neurocognitive disorders presenting with behavioral and psychological symptoms.

The primary objective of this project is to assess the feasibility and effectiveness of VR headsets with hypnotic scenarios compared with standard care in patients with ADRD presenting behavioral disturbances during hygiene care.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the St-Victor center (CHU Amiens-Picardie), including nursing home units, reinforced care units, and long-term care units;
* Patients diagnosed with ADRD presenting opposition or agitation during hygiene and toileting care;
* Affiliation to a social security scheme,
* Informed consent signed by the patient or legal representative.

Exclusion Criteria:

* Residents in terminal palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of VR headsets | up to 5 weeks
  Effectiveness of VR headsets delivering hypnotic scenarios versus standard cares in older adults with ADRD and behavioral disturbances (opposition or agitation), with the aim of reducing apprehension, pain, anxiety, and resistance during hygiene and toileting care.
  Evaluation with EPADE sclae

SECONDARY OUTCOMES:
decrease number of patients with behavioral and psychological symptoms in VR headset group | up to 5 weeks
reduced number of psychotropic drug per patient use in VR headset group | up to 5 weeks
  reduced number of psychotropic drug per patient use in VR headset group
Number of patients with improve quality of life in VH headset group | up to 5 weeks
  Number of patients with improve quality of life in VH headset group

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No